CLINICAL TRIAL: NCT05587881
Title: Clinical Study on the Impact of Covid-19 Vaccine on Safety and Efficacy of Hematological Patients Received Allogeneic Hematopoietic Sem Cell Transplantation
Brief Title: Clinical Study on the Impact of Covid-19 Vaccine on Allogeneic Hematopoietic Stem Cell Transplantation
Status: Withdrawn | Type: Observational
Why Stopped: Now, Most patients and their donor have been infected the COVID-19.
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-nCoVvaccine 01
Record Dates: First submitted 2022-10-19; First posted 2022-10-20 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2022-01

CONDITIONS: Hematologic Diseases
Keywords: Allo-HSCT; Covid-19 vaccine
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- donor with vaccine, patient without vaccine: Patients don' t receive COVID-19 vaccine before allo-HSCT but whose donors receive one dose or more doses COVID-19 vaccine(s) before stem cell collection.
  Interventions: Biological: COVID-19 vaccine(donor)
- donor without vaccine, patient with vaccine: Patients receive one dose or more doses COVID-19 vaccine(s) before allo-HSCT but whose donors don't receive COVID-19 vaccine before stem cell collection.
  Interventions: Biological: COVID-19 vaccine(donor); Biological: COVID-19 vaccine(patient)
- donor with vaccine, patient with vaccine: Patients receive one dose or more doses COVID-19 vaccine(s) before allo-HSCT and whose donors also receive one dose or more doses COVID-19 vaccine(s) before stem cell collection.
  Interventions: Biological: COVID-19 vaccine(patient)
- donor without vaccine, patient without vaccine: Patients don' t receive COVID-19 vaccine before allo-HSCT and whose donors also don't receive COVID-19 vaccine before stem cell collection.

INTERVENTIONS:
Biological: COVID-19 vaccine(donor) — Donor received COVID-19 vaccine before stem cells collection.
  Groups: donor with vaccine, patient without vaccine; donor without vaccine, patient with vaccine
Biological: COVID-19 vaccine(patient) — Patient received COVID-19 vaccine before allo-HSCT.
  Groups: donor with vaccine, patient with vaccine; donor without vaccine, patient with vaccine

SUMMARY:
Aim of this study will evaluate the Impact of Covid-19 vaccine on Safety and Efficacy of Hematological Patients Received Allogeneic Hematopoietic Stem Cell Transplantation.

DETAILED DESCRIPTION:
Since the first detection of a Corona Virus Disease 2019 (COVID-19) infection in late 2019, the syndrome coronavirus-2 (SARS-CoV-2) has spread rapidly across the globe, threatening the health and safety of an increasing number of people. The development of the SARS-CoV-2 vaccine has been shown to be effective in reducing the chance of COVID-19 infection and the severity of the disease. To control the COVID-19 pandemic, an increasing number of studies are calling for people to receive the SARS-CoV-2 vaccine, and the Chinese government is also advocating universal vaccination. However, the investigators have found in our work that as vaccination has become more widespread, clinicians have become somewhat confused about whether they can choose someone who has been vaccinated against SARS-CoV-2 as a donor for a bone marrow transplant, and what is the optimal time for allogeneic hematopoietic stem cell transplantation (allo-HSCT) in vaccined hematological patients. This study will evaluate the impact of Covid-19 vaccine on safety and efficacy of hematological patients received allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Allogeneic hematopoietic stem cell transplantation is expected to start in the short term.
2. Able and willing to provide written informed consent and comply with all requirements for study participation (including all study procedures).

Exclusion Criteria:

1. Patients or donors with a history of previous infection with SARS-Cov-2.
2. Patients or donors are currently infected with SARS-Cov-2.
3. Patients have a history of other malignancies, disease progression, or is currently on systemic therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hematological patients will receive allogeneic hematopoietic stem cell transplantation in short time.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival(PFS) | up to 12 months
  To measure the duration of response to allo-HSCT over a follow-up period of 12 months.

SECONDARY OUTCOMES:
Overall Survival(OS) | up to 12 months
  OS will be assessed from the first day of stem cells infused to death or last follow-up.
Adverse events profile | Measured 12 months after stem cells infused
  Number of participants with adverse events. Frequencies of toxicities based on NCI Common Termeinology Criteria for Adverse Events(CTCAE), version 5.0 will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D, Study Chair — The First Affilated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China